CLINICAL TRIAL: NCT03461978
Title: Ultrahigh-resolution Optical Coherence Tomography Imaging of the Anterior Eye Segment Structures - a Pilot Study
Brief Title: Ultrahigh-resolution Optical Coherence Tomography Imaging of the Anterior Eye Segment Structures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT - 010616
Record Dates: First submitted 2018-01-02; First posted 2018-03-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2022-04

CONDITIONS: Meibomian Gland Dysfunction; Cataract; Glaucoma; Corneal Transplantation; Demodicosis; Conjunctival Pathologies; Acanthamoeba Keratitis; Aniridia
MeSH Terms: conditions — Meibomian Gland Dysfunction; Cataract; Glaucoma; Acanthamoeba Keratitis; Aniridia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- 10 patients with meibomian gland dysfunction (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 10 patients with cataract (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 10 patients after minimally invasive glaucoma surgery (MIGS) (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 10 patients after partial corneal transplantation (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 5 patients with demodicosis (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 5 patients with conjunctival pathologies (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 5 patients with Acanthamoeba keratitis (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT
- 5 patients with aniridia (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT

INTERVENTIONS:
Device: Ultrahigh resolution Spectral Domain OCT — A spectrometer based ultrahigh resolution Spectral Domain OCT (SDOCT) system operating at 800 nm for the anterior chamber will be employed in the present study. The spectrum of the Ti:Sapphire laser light source is centered at 800 nm. With a full width at half maximum bandwidth of 170 nm, the axial resolution is 1.3 μm in the cornea. The transverse resolution of the employed OCT system is 21 μm at the front surface of the cornea. For measurement, patients will place their head in a modified slit lamp head rest. During the measurement period, patients will be asked to look straight forward onto an internal fixation target and to avoid blinking. Different scattering patterns, e.g. raster, circular and spiral scans will be employed.

SUMMARY:
The development of optical coherence tomography (OCT) and its application for in vivo imaging has opened entirely new opportunities in ophthalmology. The technology allows for both noninvasive visualization of the morphology and measurement of functional parameters within ocular tissues to a depth of a few millimetres even in nontransparent media. Until now the resolution of commercially available OCT systems is, however, much lower than that provided by light microscopy.

Recently, an ultrahigh-resolution OCT system was developed by our group providing resolutions of 1.7 and 17 µm in axial and lateral direction, respectively. This axial resolution is about four times better than that provided by standard OCT systems. It allows to perform in vivo imaging with a resolution close to biopsy of tissue and to visualize structures of the anterior eye segment with a remarkable richness of detail. The prototype was applied for in vivo imaging of the cornea including the precorneal tear film.

The goal of the planned pilot study is to apply this innovative imaging modality for visualization of the ultrastructure of the different parts of the anterior eye segment structures in diseased subjects, as well as in patients who underwent minimally invasive glaucoma surgery (MIGS). The obtained in vivo cross sectional images and three-dimensional data sets are hoped for contributing to the knowledge about the anatomy and physiology of the corresponding tissues. This could allow for a better interpretation of clinical features and findings obtained in slit lamp examination.

ELIGIBILITY:
Inclusion Criteria:

* For patients with meibomian gland dysfunction (MGD):

MGD as evidenced by clinical features and gland expression (MGD Grading Scheme, Appendix I (Opitz, Harthan et al. 2015))

* For cataract patients:

Cataract as evidenced from slit lamp examination, stage range between NII-NIII, CII-CIV, PII-PIII according to The Lens Opacity Classification System II (LOCS II) (Chylack, Leske et al. 1989) (Appendix II)

* For patients after minimally invasive glaucoma surgery (MIGS):

Patients with history of MIGS secondary to glaucoma

* For patients with demodicosis:

Demodicosis as evidenced from slit lamp examination and presence of Demodex confirmed by microscopic examination of the eye lashes (Liu, Sheha et al. 2010)

* For patients with conjunctival pathologies (cyst, naevus, pterygium):

Conjunctival pathologies with a clinical diagnosis of the respective

* For patients with Acanthamoeba keratitis:

Acanthamoeba keratitis as evidenced from slit lamp examination and confirmed by polymerase chain reaction (PCR) analysis of corneal epithelial and tear samples and culture isolation (Lehmann, Green et al. 1998)

* For aniridia patients:

Anirida as evidenced from slit lamp examination

Exclusion Criteria:

* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Measurement of corneal layers in ultrahigh-resolution OCT | 60 minutes
  Measurement of corneal layers in ultrahigh-resolution OCT of eyes with pathological changes in structures of the anterior eye segment.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Department of Clnical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wojtkowski M, Kaluzny B, Zawadzki RJ. New directions in ophthalmic optical coherence tomography. Optom Vis Sci. 2012 May;89(5):524-42. doi: 10.1097/OPX.0b013e31824eecb2. PMID 22446717
- [Background] Drexler W, Liu M, Kumar A, Kamali T, Unterhuber A, Leitgeb RA. Optical coherence tomography today: speed, contrast, and multimodality. J Biomed Opt. 2014;19(7):071412. doi: 10.1117/1.JBO.19.7.071412. PMID 25079820
- [Background] Werkmeister RM, Alex A, Kaya S, Unterhuber A, Hofer B, Riedl J, Bronhagl M, Vietauer M, Schmidl D, Schmoll T, Garhofer G, Drexler W, Leitgeb RA, Groeschl M, Schmetterer L. Measurement of tear film thickness using ultrahigh-resolution optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 Aug 15;54(8):5578-83. doi: 10.1167/iovs.13-11920. PMID 23847319